CLINICAL TRIAL: NCT05445661
Title: A Single Center, Double-Blinded, Split-Body, Randomized Clinical Trial of Injectable Poly-L-Lactic Acid for the Treatment of Upper Inner Arm Skin Crepiness/Laxity
Brief Title: Sculptra to Aid in Treatment of Arm Laxity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sculptra-Arms-2022-02
Record Dates: First submitted 2022-06-10; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Skin Laxity
Keywords: Skin; Volume; Volume Loss; Arms; Cosmetic
MeSH Terms: conditions — Cutis Laxa; Rhabdomyosarcoma, Alveolar | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-site, double-blinded, split-body, randomized controlled trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subject and Outcome Assessor will be unaware of which side of the subject is treated with the study device and which is treated with saline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Injectable poly-L-lactic acid (Experimental): One of the subject's arms will be treated with injectable poly-L-lactic acid (PLLA, Sculptra® Aesthetic; Galderma Laboratories; Fort Worth, TX).
  Interventions: Device: injectable poly-L-lactic acid
- Normal Saline (Sham Comparator): One of the subject's arms will be treated with injectable normal saline
  Interventions: Other: Normal Saline

INTERVENTIONS:
Device: injectable poly-L-lactic acid — Injectable biostimulant for volume loss
  Other Names: PLLA; Sculptra; Sculptra Aesthetic; Galderma
  Arms: Injectable poly-L-lactic acid
Other: Normal Saline — Sham Comparator
  Arms: Normal Saline

SUMMARY:
To assess the safety, efficacy, and patient satisfaction associated with the treatment of upper inner arm crepiness/laxity with injectable poly-L-lactic acid (PLLA, Sculptra® Aesthetic; Galderma Laboratories; Fort Worth, TX).

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to assess the safety, efficacy, and patient satisfaction associated with the treatment of upper inner arm crepiness/laxity with injectable poly-L-lactic acid (PLLA, Sculptra® Aesthetic; Galderma Laboratories; Fort Worth, TX).

Enrolled subjects will be randomized to two (2) treatment groups: "right upper medial inner arm treated" and "left upper medial inner arm treated". All subjects will receive three (3), single-sided injections of Sculptra® Aesthetic (Galderma Laboratories; Fort Worth, TX), performed one (1) month ± 7 days apart. Treatments will be provided to one side randomly assigned to either "right side" or "left side". The non-treatment side will receive bacteriostatic saline, injected in the same manner as Sculptra® Aesthetic. One (1) vial of Sculptra® Aesthetic, diluted to 16mL, will be used per treatment session.

Subjects satisfying all inclusion and no exclusion criteria will be enrolled in this trial. Prior to receiving any study treatment, mandatory digital photography with overhead lighting and VECTRA® (Canfield Scientific, Inc.; Parsippany, NJ) 3D body photography will be obtained of each subject's treatment area. In order to participate in the study, subjects must provide written informed consent to have their photographs used for research, publication, and/or commercial purposes.

ELIGIBILITY:
Inclusion Criteria:

* Adult females aged 40 to 70 years
* Subjects in good general health based on investigator's judgment and medical history
* Upper inner arm crepiness/laxity that improves when the skin of the upper inner arm is stretched or lifted superiorly
* Moderate to severe upper inner arm skin crepiness/laxity based on the Upper Inner Arm Visual Crepiness/Laxity Grading Scale (Appendix B)
* Must be willing to give and sign an informed consent form and photographic release form
* Must have a stable body weight for at least six (6) months prior to study entry
* Must be willing to maintain usual sun exposure, diet, and exercise routines for the duration of the study
* Subject agrees to avoid tanning or use of sunless tanner during the entire course of the study
* Negative urine pregnancy test result at the time of study entry (if applicable)
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

  1. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.
  2. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants, Implanon®, Depo-Provera®, double-barrier methods (e.g., condoms and spermicide), abstinence, and/or vasectomy of partner with a documented second acceptable method of birth control, should the subject become sexually active.
* Must be willing to comply with study treatments and complete the entire course of the study

Exclusion Criteria:

* Liposuction to bilateral upper arms during the 12-month period prior to study treatment or any time during the course of the study
* Mesotherapy; dermal fillers, biostimulatory injectables; radiofrequency device treatments; microfocused ultrasound device treatments; laser and light-based device treatments; microneedling; cryolipolysis; high intensity focused electromagnetic energy device treatment; or surgery (i.e., brachyplasty) during the 12-month period before study treatment
* Any investigational treatment of skin crepiness/laxity of the upper arms during the 12-month period before the study treatment
* Massage therapy during the 3-month period before study treatment.
* Creams/cosmeceuticals and/or home therapies to prevent or treat skin laxity during the four-week period before study treatment
* Subjects with scarring in the treatment areas
* History of thrombosis, post-thrombosis syndrome, or any vascular disorder of the bilateral upper extremities
* Any history of bleeding or coagulation disorders
* Subjects with tattoos or permanent implants in the treatment areas
* Subjects with a significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study
* Subjects with a history of or presence of any skin condition/disease (including but not limited to any visible rash, atopic dermatitis, psoriasis, actinic keratoses, keratinocyte carcinoma, melanoma, etc.) in the treatment area that might interfere with the diagnosis or evaluation of study parameters
* Subjects with an active bacterial, viral, or fungal infection of the treatment areas
* Subjects who spray tanned or used sunless tanners in the treatment areas four (4) weeks prior to study treatment
* History of lidocaine sensitivity deemed by the investigator to preclude the subject from enrolling into the study
* Subjects planning any cosmetic procedure to the treatment areas during the study period, other than the treatment that will be performed by the investigator
* Presence of incompletely healed wound(s) in the treatment area
* Subject who is on an immunosuppressant or has an autoimmune condition
* Female subjects who are pregnant, planning a pregnancy, or breast feeding during the study
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-20 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Upper Inner Arm Visual Skin Crepiness/Laxity Grading Scale by blinded investigator will be done to assess change. | Baseline, Day 90, Day 150, Day 240, Day 330
  Blinded Investigator will grade subjects arms at different time points using the following grading scale:
  0 None No loose skin, toned and firm skin with smooth skin surface texture
  1 Mild Mildly loose skin, somewhat toned with smooth skin surface texture
  2 Moderate Moderately loose skin, no deep tone, few wrinkles, and crepiness on skin surface
  3 Severe Very loose skin without underlying tone, multiple wrinkles and crepiness on skin surface, skin distinct from underlying subcutaneous tissue via palpation
  4 Extreme Prominent redundancy of skin without underlying tone, severe wrinkling, and crepiness on skin surface
Point of Maximal Upper Arm Skin Laxity and Circumference Measurements by blinded investigator done to assess change. | Baseline, Day 90, Day 150, Day 240, Day 330
  Blinded Investigator will take measurements of subjects arms at different time points using the following guidelines:
  Blinded Investigator Measurement of Point of Maximal Upper Arm Skin Laxity and Circumference:
  Length of Upper Arm from Axilla to Olecranon Process of Ulna Left Upper Arm Right Upper Arm cm cm
  Horizontal Distance from Axilla of Point of Maximal Upper Arm Skin Laxity Left Upper Arm Right Upper Arm cm cm
  Vertical Diameter Measured from Point of Maximal Upper Arm Laxity Left Upper Arm Right Upper Arm cm cm
  Upper Arm Circumference Measured from Point of Maximal Skin Laxity Left Upper Arm Right Upper Arm cm cm
Physician Global Aesthetic Improvement Scale (PGAIS) by blinded investigator | Day 90, Day 150, Day 240, Day 330
  Blinded Physician Global Aesthetic Improvement Scale Assessment (PGAIS) Rating Description
  1. Very Much Improved: Optimal cosmetic result in this subject.
  2. Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3. Improved: Obvious improvement in appearance from initial condition, but a re-treatment is indicated.
  4. No Change: The appearance is essentially the same as the original condition.
  5. Worse: The appearance is worse than the original condition.
  Scores write a number under each treated area or check Not Treated Left Upper Inner Arm Right Upper Inner Arm
  Not Treated Not Treated
Blinded Identification of Correct Treatment Area Photographic Assessment by blinded investigator | Day 330
  The baseline (Day 0) and 9 month (Day 330) photographs will be randomly put side-by-side and labeled either (A) or (B). The blinded investigator will then fill out the following:
  1. Do you see an improvement in the appearance of the crepiness/laxity of the upper inner arm between the two sets of photos? (Yes / No)
  2. If yes to question #1:
     1. Which is the post-treatment photograph? (A / B)
     2. Which is the treatment side? (Right / Left)

SECONDARY OUTCOMES:
Subject Global Aesthetic Improvement Scale (SGIAS) | Day 90, Day 150, Day 240, Day 330
  Subject Global Aesthetic Improvement Scale Assessment (SGAIS) How would you rate the change in appearance of your treated areas? Non-treated areas will be checked as "Not Treated" for you.
  Rating Description
  1. Very Much Improved: Optimal cosmetic result
  2. Much Improved: Marked improvement in appearance form the initial condition, but not completely optimal
  3. Improved: Obvious improvement in appearance from initial condition
  4. No Change: The appearance is essentially the same as the original condition
  5. Worse: The appearance is worse than the original condition
  Scores (write a number to rate each treated area) Left Upper Inner Arm Right Upper Inner Arm
  Not Treated Not Treated
Subject Satisfaction Questionnaire | Day 90, Day 150, Day 240, Day 330
  Subject Satisfaction Questionnaire How would you rate your satisfaction of each treated area? Non-treated areas will be checked as "Not Treated" for you.
  Rating Description 0 Not satisfied
  1. Somewhat satisfied
  2. Satisfied
  3. Very satisfied
  4. Extremely Satisfied
  Scores (write a number to rate each treated area) Left Upper Inner Arm Right Upper Inner Arm
  Not Treated Not Treated
Evaluation of side effects and adverse effects will be completed by the investigators. | Baseline, Day 30, Day 60, Day 90, Day 150, Day 240, Day 330
  Treating Investigator Evaluation of Side Effects Rating Description 0 NONE: Normal
  1. TRACE: Barely visible and localized
  2. MILD: Somewhat visible and diffuse
  3. MODERATE: Visible and diffuse
  4. SEVERE: Extremely visible and dense
  SCORES (write number under each treated area or check "Not Treated") Erythema Left Upper Inner Arm Right Upper Inner Arm
  Not Treated Not Treated
  Edema Left Upper Inner Arm Right Upper Inner Arm
  Not Treated Not Treated
  Contour Irregularity Left Upper Inner Arm Right Upper Inner Arm
  Not Treated Not Treated
  Nodules Left Upper Inner Arm Right Upper Inner Arm
  Not Treated Not Treated

IPD SHARING:
Plan to Share IPD: Undecided